CLINICAL TRIAL: NCT00619853
Title: The Influence of MCIMT (Modified Constrained Induced Movement Therapy), Bilateral Intensive Treatment, and NDT Approach on the UL Function in Children With Hemiplegic Cerebral Palsy
Acronym: CIMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-07-4624-AB-CTIL
Record Dates: First submitted 2008-02-10; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Improving the assisting hand function in children with Hemiplegic Cerebral palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: treatment approach - CIMT — CIMT, 2 months, 2Hr per day
Behavioral: treatment approach - HABIT — HABIT-2 months, 2Hr per day

SUMMARY:
The purpose of this pilot study was to compare unimanual training (CIMT) and bimanual training (HABIT) protocols aimed to improve ability of the involved hand in children with hemiplegia. Both protocols were conducted in an educational setting for 2 hours a day for 2 months, one-hour group session and one-hour individual therapy session conducted by occupational therapists or assistants.

The children in the CIMT group practiced various tasks using their involved hand with the contralateral hand constrained with a mitt. The children at the HABIT group practiced various bimanual tasks without constraint.

Twelve children (2 - 6.5 yrs.) participated in this study. The inclusion criterion included minimal extension movement of the involved wrist, and for the CIMT group, the ability to of tolerates the mitt. The children were matched in relation to cognitive level and MACS score and randomly divided into the two intervention groups.

Each child's assessment included the Quality of Upper Extremity Skills Test (QUEST), the Assisting Hand Assessment (AHA), and the Blocks and Box for children above age 5 yrs old. Range of motion (ROM) was assessed using an electronic gonimeter, and muscle tone was recorded using surface EMG and the Tardiue scale. The Child Health Questioner (CHQ) was completed by the parents before, and 6 months after, the intervention. Children were assessed starting two month before, and two month after, the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children with Hemiplegia

Exclusion Criteria:

* No ability for a minimal extension movement in the wrist

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06; Study Completion 2007-10

CONTACTS AND LOCATIONS:
Locations (1):
- MESHI kindergarten, Jerusalem, Israel